CLINICAL TRIAL: NCT04758143
Title: Most Preventable Surgical Option to Reduce Primary Spontaneous Pneumothorax Patients' Postoperative Recurrence: A Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yuka Kadomatsu (Other)
Responsible Party: Sponsor-Investigator, Yuka Kadomatsu, Subinvestigator, Nagoya University
Organization: Nagoya University (Other)
Other Study IDs: 2020-0164 20274
Record Dates: First submitted 2021-02-15; First posted 2021-02-17 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Spontaneous Pneumothorax; Recurrence; Surgery
MeSH Terms: conditions — Pneumothorax; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the most preventable option to reduce primary spontaneous postoperative recurrence.

DETAILED DESCRIPTION:
Pneumothorax is a disease in which air in the lungs leaks into the pleural cavity. It is a disease that occurs most often in young people with active social activities, and it occurs in about 100,000 people in 14 cases. The recurrence rate is as high as 17% to 54%, and the delay of the rehabilitation by the ambulatory with the treatment and prolongation of the hospitalization becomes a problem. It becomes a large failure for the youth who requires early rehabilitation. According to the latest report from the Japanese Society of Surgery, approximately 12,000 pneumothorax surgeries are performed annually in Japan. Many of them applied absorbent material to the surgical stump (coverage technique). However, there are no prospective studies, and efficacy does not appear adequately tested. It is necessary to accumulate prospective data from multiple centers to investigate the coverage technique's real effect.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have spontaneous pneumothorax diagnosed by radiography and plan to underwent initial VATS bullectomy.
2. Patients who receive informed consent to attend this study, and the agreements are provided in a document.

The consent of parents is also required, in case patients are under 20-years old.

Exclusion Criteria:

1. History of ipsilateral chest surgery.
2. Patients who only underwent exploratory surgery.
3. Patients who are judged ineligible by the investigator and the attending surgeon.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Men and Women Who Undergo Pneumothorax Surgery for the First Time at the Age of 16 to 40 Years
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of pneumothorax | within 2 years after the surgery
  Rate of ipsilateral pneumothorax recurrence detected by radiography at two years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Toyofumi Chen-Yoshikawa, PhD, Study Director — Department of Thoracic Surgery, Nagoya University Graduate Scho
Locations (1):
- Department of Thoracic Surgery, Nagoya University Graduate School of Medicine, Nagoya, Japan

REFERENCES:
- [Derived] Kadomatsu Y, Yoshioka H, Shigemitsu K, Nomata Y, Mori S, Hijiya K, Motoyama H, Ichikawa Y, Sueyoshi K, Okasaka T, Miyamoto E, Kobayashi M, Takahashi M, Fujinaga T, Takechi H, Yamagishi H, Takuwa T, Kobayashi J, Sakamoto J, Taniguchi T, Hanaoka N, Kubo Y, Chen-Yoshikawa TF. Multicentre, prospective, observational study investigating the most appropriate surgical option that can prevent the recurrence of primary spontaneous pneumothorax after surgery: the PATCH study, protocol. BMJ Open. 2021 Dec 20;11(12):e052045. doi: 10.1136/bmjopen-2021-052045. PMID 34930734